CLINICAL TRIAL: NCT04714866
Title: Cognitive Behavioral Therapy for University Students Diagnosed With Attention-deficit Hyperactivity Disorder (ADHD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Iceland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UI-HAM
Record Dates: First submitted 2021-01-08; First posted 2021-01-19 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2023-10

CONDITIONS: Attention-deficit Hyperactivity
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Cognitive behavioral therapy for ADHD
  Interventions: Behavioral: Cognitive behavioral therapy for ADHD
- waiting list group (No Intervention): No Intervention for the waiting list group

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for ADHD — CBT is a time-limited and structured approach that influences change in thoughts, feelings and behavior, leading to symptom changes.
  Arms: Interventional group

SUMMARY:
Drug treatment is often the first and only line of treatment available for ADHD. However, some do not benefit from medication. The importance of psychotherapy is becoming more widely accepted. In this study a group of university students diagnosed with ADHD will be offered cognitive behaviour therapy (CBT) in groups. The treatment will be provided by a Clinical Nurse Specialist in psychiatric nursing (CNS), in cooperation with school counsellors at the University of Iceland and the Reykjavík University. Brief CBT treatment will be offered, i.e. six group sessions, once a week over a period of six weeks.

Little is known about the effects of CBT for adults diagnosed with ADHD. The study could provide knowledge about the effects of CBT on depression, anxiety and ADHD, and on attitudes, for individuals with ADHD. The resulting knowledge might lead to improved well-being and increased quality of life.

DETAILED DESCRIPTION:
A treatment manual for adults with ADHD was written based on the CBT model described in Young and Bramham's Handbook on ADHD in Adults (2007), Greenberger and Padesky's Mind Over Mood (2016) and Honos-Webb's The Gift of Adult ADD (2008). Emphasis will be on collaboration, incentive, group interaction and therapy rather than didactic instruction. The manual-based group treatment will be conducted in six sessions. An web page was developed in collaboration with the Faculty of Electrical and Computer Engineering at the University of Iceland containing homework and coping skills assignments to support the participants during therapy. A pilot study has been conducted where adults (n= 5) previously diagnosed with ADHD was offered group CBT in six sessions. The usefulness and benefits of the manual and the App will be evaluated by using questionnaires. Participants was also asked about the group format. The manual and the App will be further developed in light of the pilot study's results.

University students with ADHD (n= ........) previously diagnosed by a psychiatrist or a psychologist, will be offered group CBT in six sessions. The study will be introduced to the university students by the school counsellors at the University of Iceland and Reykjavik University. The school counsellors will contact the students and offer them to take part in the therapy. Participants will be randomized into two groups: a waiting list group and a therapy group. The waiting list group will subsequently be offered treatment after a wait of approximately six months. The therapy will be provided by a CNS. CBT sessions will take place once a week over a period of six weeks.

Assessments will be conducted before the intervention (baseline), at end of treatment, and at six-month follow-up. In addition, half of the participants will be placed on a waiting list, and will be assessed at the same time as the intervention group (baseline) and again six weeks later, and again six month after that, and will serve as a waiting list comparison group. They will subsequently be offered the treatment intervention and will be included in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

University students who have previously been diagnosed with ADHD, and are fluent in Icelandic. Students with co-morbid disorders such as dyslexia, anxiety or depression will be included. Students currently receiving other psychological or medical treatment will be included.

Exclusion Criteria:

Students with psychotic disorders, autism spectrum disorders or drug dependence will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Beck´s Depression Inventory II | T1 (at baseline)
  The inventory includes 21 items that measure depression and well-being during the past two weeks. Options range from 0-3 in each item. The scores can range between 0 and 63. α = 0.89 - 0.94
Beck´s Depression Inventory II | T2 (post-treatment after 6 weeks)
  The inventory includes 21 items that measure depression and well-being during the past two weeks. Options range from 0-3 in each item. The scores can range between 0 and 63. α = 0.89 - 0.94
Beck´s Depression Inventory II | T3 (follow-up 4-6 months post treatment)
  The inventory includes 21 items that measure depression and well-being during the past two weeks. Options range from 0-3 in each item. The scores can range between 0 and 63. α = 0.89 - 0.94
Sense of coherence | T1 (at baseline)
  A. Antonovsky, The inventory includes 29- items with three components; Comprehensibility, manageability and meaningfulness. The items are measured on a 7-point scale. Cronbach´s alpha 0.70-0.95
Sense of coherence | T2 (post-treatment after 6 weeks)
  A. Antonovsky, The inventory includes 29- items with three components; Comprehensibility, manageability and meaningfulness. The items are measured on a 7-point scale. Cronbach´s alpha 0.70-0.95
Sense of coherence | T3 (follow-up 4-6 months post treatment)
  A. Antonovsky, The inventory includes 29- items with three components; Comprehensibility, manageability and meaningfulness. The items are measured on a 7-point scale. Cronbach´s alpha 0.70-0.95
Well-being | T1 (at baseline)
  Dupuy, the questionnaire measures well-being and to how they feel about their inner personal state. The inventory includes 18 items that include negative and positive questions with six components; anxiety, depression, general health, positive well-being, self-control and vitality. Cronbac´s alpha 0.91-0.94
Well-being | T2 (post-treatment after 6 weeks)
  Dupuy, the questionnaire measures well-being and to how they feel about their inner personal state. The inventory includes 18 items that include negative and positive questions with six components; anxiety, depression, general health, positive well-being, self-control and vitality. Cronbac´s alpha 0.91-0.94
Well-being | T3 (follow-up 4-6 months post treatment)
  Dupuy, the questionnaire measures well-being and to how they feel about their inner personal state. The inventory includes 18 items that include negative and positive questions with six components; anxiety, depression, general health, positive well-being, self-control and vitality. Cronbac´s alpha 0.91-0.94
Barkley Adult ADHD rating Scale | T1 (at baseline)
  The questionnaire includes 18- items that are based on DSM-IV criteria for ADHD and is evaluated on a 4-point Likert scale. Cronbach's alpha 0.91-0.93 in the Icelandic version
Barkley Adult ADHD rating Scale | T2 (post-treatment after 6 weeks)
  The questionnaire includes 18- items that are based on DSM-IV criteria for ADHD and is evaluated on a 4-point Likert scale. Cronbach's alpha 0.91-0.93 in the Icelandic version
Barkley Adult ADHD rating Scale | T3 (follow-up 4-6 months post treatment)
  The questionnaire includes 18- items that are based on DSM-IV criteria for ADHD and is evaluated on a 4-point Likert scale. Cronbach's alpha 0.91-0.93 in the Icelandic version
Rosenberg Self-Esteem Scale | T1 (at baseline)
  The scale is a 10-item scale that measures global self-worth using a 4-point Likert scale. Cronbach's alpha 0.87-0.93
Rosenberg Self-Esteem Scale | T2 (post-treatment after 6 weeks)
  The scale is a 10-item scale that measures global self-worth using a 4-point Likert scale. Cronbach's alpha 0.87-0.93
Rosenberg Self-Esteem Scale | T3 (follow-up 4-6 months post treatment)
  The scale is a 10-item scale that measures global self-worth using a 4-point Likert scale. Cronbach's alpha 0.87-0.93
SCL-90 Anxiety subscale | T1 (at baseline)
  The questionnaire includes 10 items related to anxiety symptoms that are evaluated on a 5-point Likert scale. Cronbach's alpha 0.90
SCL-90 Anxiety subscale | T2 (post-treatment after 6 weeks)
  The questionnaire includes 10 items related to anxiety symptoms that are evaluated on a 5-point Likert scale. Cronbach's alpha 0.90
SCL-90 Anxiety subscale | T3 (follow-up 4-6 months post treatment)
  The questionnaire includes 10 items related to anxiety symptoms that are evaluated on a 5-point Likert scale. Cronbach's alpha 0.90
Automatic Thoughts Questionnaire | T1 (at baseline)
  The scale includes 30-item self-statements that measures the frequency of automatic negative thoughts. Thoughts are evaluated on a 5-point scale, how frequent the thoughts are. Chroma's alpha=0.96
Automatic Thoughts Questionnaire | T2 (post-treatment after 6 weeks)
  The scale includes 30-item self-statements that measures the frequency of automatic negative thoughts. Thoughts are evaluated on a 5-point scale, how frequent the thoughts are. Chroma's alpha=0.96
Automatic Thoughts Questionnaire | T3 (follow-up 4-6 months post treatment)
  The scale includes 30-item self-statements that measures the frequency of automatic negative thoughts. Thoughts are evaluated on a 5-point scale, how frequent the thoughts are. Chroma's alpha=0.96

CONTACTS AND LOCATIONS:
Overall Officials: Erla K Svavarsdottir, PhD, Study Director — University of Iceland
Locations (1):
- University of Iceland, Reykjavik, Sæmundargata 2, Iceland

IPD SHARING:
Plan to Share IPD: No